CLINICAL TRIAL: NCT07369089
Title: KETAMORE: TARGETING TREATMENT-RESISTANT OUD WITH KETAMINE-ASSISTED MINDFULNESS-ORIENTED RECOVERY ENHANCEMENT
Brief Title: Targeting Treatment-Resistant OUD With Ketamine-Assisted Mindfulness Oriented Recovery Enhancement
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Garland, Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 177164
Record Dates: First submitted 2026-01-23; First posted 2026-01-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
Keywords: Mindfulness; Ketamine; Opioid Use disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Ketamine; Self-Help Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine-Assisted Psychotherapy Plus Mindfulness-Oriented Recovery Enhancement (KetaMORE) (Experimental): Participants assigned to this arm will receive ketamine-assisted psychotherapy combined with Mindfulness-Oriented Recovery Enhancement (MORE). MORE is delivered as a structured, manualized behavioral intervention designed to reduce opioid use by targeting craving, negative affect, and maladaptive reward processing through mindfulness training, cognitive reappraisal, and savoring techniques.
  Interventions: Drug: Ketamine; Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE)
- Ketamine-Assisted Psychotherapy Plus Support Group (Active Comparator): Participants assigned to this arm will receive ketamine-assisted psychotherapy combined with a support group intervention. The support group provides nonspecific therapeutic support and group discussion but does not include mindfulness training or structured skills from Mindfulness-Oriented Recovery Enhancement.
  Interventions: Drug: Ketamine; Behavioral: Support Group

INTERVENTIONS:
Drug: Ketamine — Ketamine will be administered as part of ketamine-assisted psychotherapy under medical supervision according to the study protocol. Ketamine dosing and administration procedures will be identical across study arms.
Behavioral: Mindfulness-Oriented Recovery Enhancement (MORE) — Mindfulness-Oriented Recovery Enhancement is a manualized, evidence-based intervention integrating mindfulness practices, cognitive reappraisal, and savoring exercises to reduce craving, improve emotional regulation, and support recovery from opioid use disorder. MORE sessions are delivered in a group format and coordinated with ketamine-assisted psychotherapy sessions.
  Arms: Ketamine-Assisted Psychotherapy Plus Mindfulness-Oriented Recovery Enhancement (KetaMORE)
Behavioral: Support Group — The support group intervention consists of therapist-led group sessions focused on emotional support and discussion of recovery-related experiences. This condition is designed to match the MORE intervention in duration and therapist contact while excluding mindfulness-based or structured skills training.
  Arms: Ketamine-Assisted Psychotherapy Plus Support Group

SUMMARY:
The goal of this clinical trial is to examine the usefulness of Mindfulness-Oriented Recovery Enhancement combined with Ketamine-Assisted Psychotherapy (KetaMORE) for individuals with opioid use disorder who are receiving medication treatment. The main question it aims to answer is whether individuals with opioid use disorder who receive Mindfulness-Oriented Recovery Enhancement in combination with Ketamine-Assisted Psychotherapy will demonstrate greater reductions in opioid use and craving than individuals who receive Ketamine-Assisted Psychotherapy with a non-mindfulness support group.

Participants will be randomly assigned to receive either Mindfulness-Oriented Recovery Enhancement combined with Ketamine-Assisted Psychotherapy or Ketamine-Assisted Psychotherapy combined with a support group control condition. Researchers will compare these groups on days of opioid use, time to first opioid use lapse, craving, and mood, assessed using ecological momentary assessments and standardized measures collected during treatment and follow-up.

DETAILED DESCRIPTION:
This study is a Phase II, two-arm, parallel randomized controlled trial designed to evaluate the efficacy of Mindfulness-Oriented Recovery Enhancement combined with Ketamine-Assisted Psychotherapy (KetaMORE) compared to Ketamine-Assisted Psychotherapy paired with a support group control condition for individuals with opioid use disorder receiving medications for opioid use disorder (MOUD), including buprenorphine.

Participants will be randomized in a 1:1 ratio to one of two conditions: (1) Ketamine-Assisted Psychotherapy combined with Mindfulness-Oriented Recovery Enhancement, or (2) Ketamine-Assisted Psychotherapy combined with a support group providing nonspecific therapeutic support without mindfulness training. Both groups will receive identical ketamine dosing and psychotherapy components; the conditions will differ only in the adjunctive behavioral intervention.

Mindfulness-Oriented Recovery Enhancement is a manualized, evidence-based intervention integrating mindfulness training, cognitive reappraisal, and savoring techniques to reduce craving, negative affect, and maladaptive reward processing associated with substance use. The support group control condition is designed to match therapist contact and group support while excluding mindfulness-based content.

Participants will complete assessments at baseline, during treatment, post-treatment, and follow-up. Primary outcomes will include number of days of opioid use and time to first opioid use lapse. Secondary outcomes will include opioid craving and mood symptoms. Ecological momentary assessments will be used to capture daily fluctuations in substance use, craving, and affect throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking .
2. DSM-5 criteria for Opioid Use Disorder (OUD).
3. Documented evidence (by urine toxicology) of current illicit drug use (upon screening) or by self-report on the Addiction Severity Index (ASI).
4. Men/Women >/= 18
5. Current prescription of a buprenorphine-containing product.
6. Have a support person that would be able to escort the subject home on the evening of the ketamine dosing session. The use of ride services will not be permitted (e.g., Uber, Lift, taxi, etc.).
7. Agreement to adhere to Lifestyle Considerations

Exclusion Criteria:

* 1. A primary DSM-5 Axis I diagnosis of schizophrenia, schizoaffective disorder, dissociative identity disorder, or bipolar I/II disorder as determined by psychiatric evaluation.

  2. Has baseline hypertension (≥160 SBP or ≥100 DBP), after repeated measurements. Note: Participants with hypertension that has been controlled by medication down to <160 Systolic blood pressure (SBP) and <100 diastolic blood pressure (DBP) will be allowed participate.

  3. Has baseline abnormal resting heart rate (>100 or <60). 4. History of cardiovascular disease, including but not limited to clinically significant coronary artery disease, cardiac hypertrophy, cardiac ischemia, congestive heart failure, myocardial infarction, angina pectoris, coronary artery bypass graft or artificial heart valve, stroke, transient ischemic attack, or any clinically significant arrhythmia.

  5. Has QTcf >450msec for men or women on EKG. Note: Participants may qualify for the study if QTc 450-480 msec on one EKG, but then <=450 msec on repeat EKG. If QT-prolonging medications are started or increased in dose after enrollment and prior to ketamine administration, a repeat EKG must be done >12-hours after this change in order to assure continued safe enrollment in the trial.

  6. Active suicidal intent or suicidal or non-suicidal self-injurious behaviors, as defined by a "yes" response to question 4 on C-SSRS within the past 6 months at screening or prior to dosing (Active Suicidal Ideation with Some Intent to Act, with or without Specific Plan).

  7. Suicidal behaviors within the last 6 month. 8. History of allergy or hypersensitivity reaction to ketamine. 9. History of ketamine use disorder. 10. History of intracranial bleeding or stroke. 11. Current intracranial mass. 12. Seizure within the last 6 months prior to screening visit. 13. Baseline oxygen saturation <95%. 14. Current significant liver disease. 15. Meets the following laboratory parameters:
  1. Any significant liver diseases or symptoms of liver disease regardless of liver enzyme levels.
  2. Asymptomatic alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >=5x upper limit of normal (ULN).
  3. Symptomatic ALT or AST >= 2x ULN.
  4. AST/ALT >3 upper limit of normal (ULN)
  5. Total bilirubin > 1.5x ULN (Gilbert syndrome is allowed).
  6. Alkaline phosphatase (ALP) >2x ULN.
  7. Renal insufficiency (i.e., estimated glomerular filtration rate (eGFR) < 30 milliliter/minute (mL/min) /1.73 m^2 (using the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation), Creatinine Clearance (CrCl) < 30 mL/min (using the Cockcroft-Gault Equation), or current dialysis)).

     16. Currently pregnant or breastfeeding. 17. Has uncontrolled insulin-dependent diabetes and has had a hospitalization for diabetes-related complication within 6 months of signing ICF.

     18. Diagnosed cognitive impairments, including dementia, mild cognitive impairment, traumatic brain injury, or developmental delays, that would prevent the participant from completing the study protocol, as identified by self-disclosure when asked in eligibility screening question.

     19. Individuals prescribed monoamine oxidase inhibitors.(see Appendix 1) 20. Individuals prescribed medications that are CYP2B6 inhibitors or inducers (see Appendix 1) 21. Patients taking >2 mg of lorazepam-equivalents per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Abstinence | From day 15 through 84.
  Abstinence as measured by timeline followback and triangulated by drug screen.

SECONDARY OUTCOMES:
MOUD discontinuation | From day 15 to 84.
  Discontinuation of medications for opioid use disorder (MOUD), defined as cessation of prescribed MOUD during the study period using the Timeline Follow-back and biochemically verified use via drug screens.
Opioid Craving (Ecological Momentary Assessments) | From baseline through week 12.
  Opioid craving assessed using ecological momentary assessment (EMA) on a 0-10 numeric rating scale (0=no craving, 10 extreme craving).
Opioid Craving (Desires for Drug Questionnaire) | From baseline to week 12.
  Opioid craving measured using the Desires for Drug Questionnaire (DDQ), a validated self-report measure of desire and urge to use opioids (0= Strongly Disagree, 6= Strongly Agree)
Quality of life (WHO-5) | From baseline to week 12.
  Quality of life assessed using the World Health Organization Five Well-Being Index (WHO-5), a brief measure of subjective psychological well-being. (0= At no time, 5= All of the time)
Depressive Symptoms (Patient Health Questionnaire-9) | From baseline to week 12.
  Depressive symptom severity assessed using the Patient Health Questionnaire-9 (PHQ-9). (0= Not at all, 3= Nearly every day)
Post-Traumatic Stress Symptoms (PTSD Checklist for DSM-5) | From baseline to week 12.
  Post-traumatic stress symptom severity assessed using the PTSD Checklist for DSM-5 (PCL-5). (0 = Not at all, 4= Extremely )
Anhedonia (Snaith-Hamilton Pleasure Scale) | From baseline to week 12.
  Anhedonia assessed using the Snaith-Hamilton Pleasure Scale (SHAPS), a validated measure of reduced capacity to experience pleasure. (1=Strongly Disagree, 4= Strongly Agree)
Psychological Distress (Depression Anxiety Stress Scales) | From baseline to week 12.
  Psychological distress assessed using the Depression Anxiety Stress Scales (DASS). (0= Did not apply to me at all, 3= Applied to me very much or most of the time)
Positive and Negative Affect (Positive and Negative Affect Schedule) | From baseline to week 12.
  Positive and negative affect assessed using the Positive and Negative Affect Schedule (PANAS). (1= Very slightly or not at all, 5= Extremely)
Pain (PEG Scale) | Baseline to week 12.
  Pain severity and pain-related interference assessed using the PEG scale. (0= no pain or interference, 10= Worst imaginable pain or interference)
Momentary affective state | Baseline through week 12.
  Momentary affective state measured by EMA on 0-10 numeric rating scale (0=low affect, 10=high affect).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - University Of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
De-Identified participant data will be shared for approved purposes with assigned data access agreement (i.e., meta-analysis)
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after publication of the primary, secondary, and mechanistic outcomes of the trial.
Access Criteria: Data will be available with a signed data access agreement